CLINICAL TRIAL: NCT00422903
Title: Letrozole Versus Letrozole Plus Lapatinib (GW572016) in Hormone-sensitive, HER-2 Negative Operable Breast Cancer. A Double Blind Randomized Phase II Study With Biomarker Evaluation.
Brief Title: Letrozole In Combination With Lapatinib In Neoadjuvant Treatment Of Early Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EGF107692
Record Dates: First submitted 2007-01-16; First posted 2007-01-17 (Estimated); Results first posted 2012-08-29 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-03

CONDITIONS: Neoplasms, Breast
Keywords: neo-adjuvant; letrozole; lapatinib; primary breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Letrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Letrozole plus placebo (Placebo Comparator): Letrozole 2.5 mg administered orally fro 6 mos. plus placebo 1500 mg administered orally throughout the study until definitive surgery
  Interventions: Drug: letrozole; Other: placebo
- Letrozole plus lapatininb (Experimental): Letrozole 2.5 mg administered orally fro 6 mos. plus lapatinib 1500 mg administered orally throughout the study until definitive surgery
  Interventions: Drug: lapatinib; Drug: letrozole

INTERVENTIONS:
Drug: lapatinib — 1500 mg administered orally daily
  Arms: Letrozole plus lapatininb
Drug: letrozole — 2.5 mg administered orally daily
Other: placebo — 1500 mg administered orally daily
  Arms: Letrozole plus placebo

SUMMARY:
Evaluate the percentage of clinical objective responses (cOR) in patients with HER2 negative early breast cancer treated with pre operative (neoadjuvant)lapatinib and letrozole

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed infiltrating primary breast cancer of 2.0 cm or more in largest clinical diameter
* ER and/or PgR positive cancer (> 10% of positive cancer cell assessed by IHC)
* Postmenopausal status, defined by at least one of the following:

  ≥ 60 years of age < 60 years of age and amenorrheic for ≥ 12 months prior to day 1 < 60 years of age and amenorrheic for < 12 months prior to day, or without a uterus: luteinizing hormone (LH) and follicle stimulating hormone (FSH) values within postmenopausal range Prior bilateral oophorectomy Prior radiation castration with amenorrhea for at least 6 months
* HER2 negative tumors (IHC 0-2+, or FISH negative)
* Availability of tumor tissue suitable for biological and molecular examination before starting primary treatment
* Age over 18 years
* ECOG PS 0-1
* Normal organ and marrow function as defined below:

leukocytes > 3000/mL absolute neutrophil count > 1,500/mL platelets > 100,000/mL total bilirubin within normal institutional limits AST (SGOT)/ALT(SGPT)< 2.5 X institutional upper limit of normal Creatinine within normal institutional limits

* Cardiac ejection fraction within the institutional range of normal as measured by echocardiogram or MUGA scan.
* Eligibility of patients receiving medications or substances known to affect, or with the potential to affect the activity or pharmacokinetics of lapatinib will be determined following review of their use by the Principal Investigator.

A list of medications and substances known or with the potential to interact with CYP450 isoenzymes is provided

* Ability to understand and the willingness to sign a written informed consent document.
* Ability to swallow and retain oral medication.

Exclusion criteria:

* Stage IIIB, IIIC, and inflammatory breast cancer
* Stage IV breast cancer
* Contraindication to the treatment with letrozole
* Prior treatment with chemotherapy, endocrine therapy or radiotherapy. Prior treatment with EGFR targeting therapies
* Treatment with any other investigational agents, or with all herbal (alternative) medicines
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lapatinib
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* HIV-positive patients receiving combination anti-retroviral therapy
* GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis)
* Concomitant requirement for medication classified as CYP3A4 inducers or inhibitors (See section 3.7.4.2 Other concomitant treatments)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2007-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- Italy (13):
  - GSK Investigational Site, Brindisi, Apulia
  - GSK Investigational Site, Carpi (MO), Emilia-Romagna
  - GSK Investigational Site, Forlì, Emilia-Romagna
  - GSK Investigational Site, Modena, Emilia-Romagna
  - GSK Investigational Site, Piacenza, Emilia-Romagna
  - GSK Investigational Site, Rimini, Emilia-Romagna
  - GSK Investigational Site, Treviglio (BG), Lombardy
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, Chieti
  - GSK Investigational Site, Cremona
  - GSK Investigational Site, Perugia
  - GSK Investigational Site, Reggio Emilia
  - GSK Investigational Site, Varese
- GSK Investigational Site, Badalona, Spain

RESULTS

PARTICIPANT FLOW:
Groups:
- Letrozole + Placebo: Letrozole tablets in the dose of 2.5 milligrams (mg) plus matching placebo were administered orally once daily for 6 months prior to surgery.
- Letrozole + Lapatinib: Letrozole tablets in the dose of 2.5 mg plus lapatinib ditosylate monohydrate tablets in the dose of 1500 mg were administered orally once daily for 6 months prior to surgery.
Period: Overall Study
Arm/Group | Letrozole + Placebo | Letrozole + Lapatinib
Started | 49 | 43
Completed | 45 | 38
Not Completed | 4 | 5
Not completed — Disease Progression | 3 | 1
Not completed — Adverse Event | 0 | 2
Not completed — Informed Consent Withdrawn | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Letrozole + Placebo | Letrozole + Lapatinib | Total
Number analyzed (Participants) | 49 | 43 | 92
Age, Continuous [Median (Full Range); unit: Years] | 70 [47 to 88] | 70 [49 to 88] | 70 [47 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 43 | 92
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Objective Response (cOR) in the Breast, Evaluated by an Independent Radiological Evaluation Monitoring Committee
Description: cOR is defined as the documented evidence of complete response (CR) and partial response (PR) as assessed by ultrasound examination using Response Evaluation Criteria In Solid Tumors (RECIST). CR is defined as the disappearance of all target lesions (TLs) and non-TLs and the appearance of no new lesions (NLs). PR for TLs is defined as a >=30% decrease in the sum of the longest diameter (LD) of TLs, taking as a reference the Baseline sum LD. For non-TLs, it is defined as the persistence of >=1 non-TL and no new TLs or non-TLs.
Time Frame: From Baseline (Day 1) up to 6 months, evaluated every 12 weeks
Population: Intent-to-Treat (ITT) Population: all participants who entered the study and received at least one dose of letrozole. Three participants withdrew consent and were not included in the efficacy analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Letrozole + Placebo | Letrozole + Lapatinib
Number analyzed (Participants) | 48 | 41
percentage of participants
  CR | 2 | 12
  PR | 58 | 54

2. Primary Outcome: Percentage of Participants With Various Responses in the Breast, Evaluated Using Per Protocol Criteria
Description: Complete clinical response=nodule not detectable; all ultrasound abnormalities detected at diagnosis have disappeared. Partial clinical response=the tumor's longest diameter (LD) is reduced by 50% or more; ultrasound characteristics of the tumor persist. Minimal response=the tumor's LD is reduced by 25%-49%. Stable disease=the tumor's LD is decreased by less than 25% and is increased by no more than 25% from the starting value. Progressive disease=the tumor's LD is increased by more than 25% from the starting value. Participants who were not evaluable did not have data available.
Time Frame: From Baseline (Day 1) up to 6 months, evaluated every 12 weeks
Population: ITT Population. Three participants withdrew consent and were not included in the efficacy analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Letrozole + Placebo | Letrozole + Lapatinib
Number analyzed (Participants) | 48 | 41
percentage of participants
  Complete Response | 2 | 12
  Partial Response | 27 | 34
  Minimal Response | 40 | 24
  Stable Disease | 33 | 20
  Progressive Disease | 6 | 2
  Not Evaluable | 2 | 7

3. Secondary Outcome: Percentage of Participants With Pathological Complete Response (pCR) in the Breast and Axillary Nodes, Evaluated Using Miller and Payne Criteria
Description: pCR is defined as the complete absence of infiltrating tumor cells (TCs) in the breast and lymph nodes. Miller and Payne criteria: Grade 1, no change/some alteration to individual malignant cells, but no reduction in overall cellularity; Grade 2, up to a 30% loss in TCs; Grade 3, between an estimated 30% and 90% reduction in TCs; Grade 4, more than a 90% reduction in TCs, only small cluster/dispersed cells remaining; Grade 5, no malignant identifiable cells; carcinoma in the milk ducts may be present. Grades 1 and 2 = No response; Grades 3 and 4= PR; Grade 5 = CR.
Time Frame: At the point of definitive surgery (up to 6 months after Baseline)
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Letrozole + Placebo | Letrozole + Lapatinib
Number analyzed (Participants) | 49 | 43
Percentage of participants | 0 [0.0 to 7.3] | 0 [0.0 to 8.2]

4. Secondary Outcome: Number of Participants With Breast Tumors Per Pathological Stage at Surgery
Description: Tumors were categorized as follows: T0, no evidence of primary tumor, but carcinoma of the milk ducts, accumulation of abnormal cells in the breast lobules, or Paget disease (cancer condition that appears like a skin disease involving the breast nipple) with no associated tumor mass; T1, tumor was <=2 centimeters (cm) across; T2, tumor was >2 cm but <5 cm across; T3, tumor was >5 cm across; T4, tumor of any size growing into the chest wall or skin, including inflammatory breast cancer.
Time Frame: At the point of definitive surgery (up to 6 months after Baseline)
Population: ITT Population. Only those participants contributing data were analyzed.
Measure: Number; unit: participants
Arm/Group | Letrozole + Placebo | Letrozole + Lapatinib
Number analyzed (Participants) | 47 | 42
participants
  T0 | 1 | 0
  T1 | 20 | 26
  T2 | 24 | 12
  T3 | 2 | 2
  T4 | 0 | 2

5. Secondary Outcome: Number of Participants With the Indicated Nodal Status at Surgery
Description: The nodal status of cancer indicates the involvement of lymph nodes in the participant with cancer. N0 indicates no involvement of lymph nodes, and N+ indicates involvement of lymph nodes.
Time Frame: At the point of definitive surgery (up to 6 months after Baseline)
Population: ITT Population. Only those participants contributing data were analyzed.
Measure: Number; unit: participants
Arm/Group | Letrozole + Placebo | Letrozole + Lapatinib
Number analyzed (Participants) | 47 | 42
participants
  N0 | 19 | 21
  N+ | 28 | 21

6. Secondary Outcome: Number of Participants With the Indicated Type of Surgery
Description: Mastectomy is the medical term for the surgical removal of one or both breasts. Breast-conserving surgery (BCS) involves removing only the affected part of the breast tissue during surgery, as opposed to removal of the entire breast.
Time Frame: At the point of definitive surgery (up to 6 months after Baseline 1)
Population: ITT Population. Only those participants contributing data were analyzed.
Measure: Number; unit: participants
Arm/Group | Letrozole + Placebo | Letrozole + Lapatinib
Number analyzed (Participants) | 49 | 43
participants
  Mastectomy | 13 | 15
  BCS | 34 | 27
  Not done | 2 | 1

7. Secondary Outcome: Percentage of Participants With Conversion From Planned Mastectomy at Baseline to BCS at Surgery
Description: The percentage of participants who were planned to undergo a mastectomy at baseline but later underwent BCS was measured.
Time Frame: At the point of definitive surgery (up to 6 months after Baseline)
Population: ITT Population. Only those participants contributing data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Letrozole + Placebo | Letrozole + Lapatinib
Number analyzed (Participants) | 49 | 43
percentage of participants | 56 | 46

8. Secondary Outcome: Number of Participants With the Indicated Adverse Events With a Classification of >=Grade 2
Description: Toxicity was measured in grades (severity of the AE) as per National Cancer Institute Common Toxicity Criteria for Adverse Event (NCI CTCAE) version (v) 3.0. The CTCAE v3.0 displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1, mild; Grade 2, moderate; Grade 3, severe; Grade 4, life-threatening/disabling; Grade 5, death related to the AE. Mucositis is the painful inflammation and ulceration of the mucous membranes lining the digestive tract, and hypertension is high blood pressure.
Time Frame: From Baseline (Day 1) up to 6 months (until definitive surgery)
Population: ITT Population. Only those participants contributing data were analyzed.
Measure: Number; unit: participants
Arm/Group | Letrozole + Placebo | Letrozole + Lapatinib
Number analyzed (Participants) | 49 | 43
participants
  Musculoskeletal pain | 4 | 2
  Diarrhea | 2 | 10
  Mucositis | 0 | 8
  Liver toxicity | 1 | 4
  Skin disorders | 1 | 18
  Hypertension | 1 | 2

9. Secondary Outcome: Mean Left Ventricular Ejection Fraction (LVEF)
Description: Cardiac safety was evaluated as any signs or symptoms of deterioration in LVEF. LVEF is the measurement of how much blood is being pumped out of the left ventricle of the heart (the main pumping chamber) with each contraction. LVEF was evaluated using NCI CTCAE.
Time Frame: Baseline (Day 1), after 12 weeks, and after 24 weeks
Population: ITT Population. Only those participants contributing data were analyzed.
Measure: Mean (Full Range); unit: Percent volume
Arm/Group | Letrozole + Placebo | Letrozole + Lapatinib
Number analyzed (Participants) | 49 | 43
Percent volume
  Baseline | 61 [50 to 78] | 61 [54 to 76]
  After 12 weeks | 62 [50 to 76] | 60 [52 to 75]
  After 24 weeks | 61 [50 to 84] | 59 [50 to 75]

10. Secondary Outcome: Time to Treatment Failure From the Start of the Primary Therapy
Description: Time to treatment failure is calculated as the interval between the date of randomization and the occurrence of local tumor progression (including ipsilateral [on the same side] and controlateral breast tumor progression), distant tumor progression, permanent treatment discontinuation (either for the experimental or conventional treatment arm), or death for any cause.
Time Frame: From Baseline (Day 1) up to study withdrawal (approx. 66 months)
Population: ITT Population. Only those participants contributing data were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Letrozole + Placebo | Letrozole + Lapatinib
Number analyzed (Participants) | 13 | 6
Months | 32.2 [6.3 to 38.5] | 22.2 [NA to NA] — The confidence limits for the median value are not estimable because there are no time points that satisfy the condition using the method of Klein and Moeschberger (1997).

ADVERSE EVENTS:
Arm/Group | Letrozole + Placebo | Letrozole + Lapatinib
Serious Adverse Events (participants affected / at risk) | 1/49 | 3/43
Other Adverse Events (participants affected / at risk) | 20/49 | 36/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Letrozole + Placebo (N=49) | Letrozole + Lapatinib (N=43)
Myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Sphincter of Oddi dysfunction (Hepatobiliary disorders) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Letrozole + Placebo (N=49) | Letrozole + Lapatinib (N=43)
Astenia/Fatigue (General disorders) | 6 | 7
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 0 | 25
Diarrhea (Gastrointestinal disorders) | 5 | 26
Dyspepsia (Gastrointestinal disorders) | 5 | 5
LFT transaminases (Investigations) | 0 | 8
Mucositis (Injury, poisoning and procedural complications) | 0 | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 | 6
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 5
Nausea (Gastrointestinal disorders) | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.